CLINICAL TRIAL: NCT05546281
Title: Study of the Characteristics of Orthorexia Nervosa in the Population Living with Type 1 Diabetes
Acronym: Santal-DT1
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Sylvain Iceta, Principal Investigator - Assitant Professor, Laval University
Other Study IDs: 2023-3914, 22258
Record Dates: First submitted 2022-09-16; First posted 2022-09-19 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes; Orthorexia nervosa; Eating Disorder; Mental Health
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Orthorexia Nervosa; Feeding and Eating Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
In the general population, the excessive and constant desire to control one's diet and body has become increasingly problematic. Indeed, the demand for control over one's diet and body is now an unspoken social prescription that can lead in some cases to eating disorders. In patients with type 1 diabetes (T1D), these concerns are even more central, as they are accentuated by the very nature of the treatment of the disease (dietary modification, insulin compensation according to food intake, etc.). Studies on adolescents with T1D show that the prevalence of eating disorders would be present in at least 1 in 5 patients. Among these disorders, orthorexia is of particular interest. Indeed, orthorexia was defined in 1997 by Steven Bratman as a rigid eating behavior based on the avoidance of foods considered qualitatively unhealthy. More precisely, orthorexia is characterized by a constant preoccupation with one's diet and persistent nutritional (or health) beliefs that take precedence over food pleasure. It has been estimated that the prevalence of orthorexia in patients living with T1D may be as high as 80%. We are currently conducting a study on the mechanisms of orthorexia in the general population of Quebec (the results of phase 1 of this study are being analyzed). We now wish to conduct the same study in a population with T1D, which has a higher prevalence of people with orthorexia nervosa.

The main objective of this study is to investigate the characteristics of orthorexia nervosa (obsessions and fixations on healthy eating) in the Quebec population with T1D from the BETTER Registry.

DETAILED DESCRIPTION:
The BETTER registry is supervised by Dr. Rabasa-Lhoret and Dr. Brazeau and co-funded by CIHR and JDRF: more than 2000 patients with T1D are currently in the registry, of which 98% of the participants have agreed to be contacted for future research studies. This will be done by comparing food categorization strategies between control subjects from the previous study (results under analysis) and subjects with orthorexia nervosa traits in the T1D patient population, and also by testing the hypothesis of dysfunctions specific to the orthorexia population of executive functions (including attention, cognitive flexibility, inhibition and working memory) in the general domain and then more specifically in the food domain.

Considering the existing literature on orthorexia described above, and in particular the definition of orthorexia nervosa (orthorexia nervosa is defined as obsessions and fixations on healthy eating leading to negative emotional and behavioral consequences for the individual, e.g., excessive anxiety, social isolation), as well as the strong correlations observed in the literature between distress, anxiety, and diabetes, the hypotheses are the following:

* Hypothesis 1: The more orthorexic traits subjects exhibit, the more quickly they categorize foods into healthy/unhealthy.
* Hypothesis 2: The likelihood that a food, regardless of its properties, will be categorized as unhealthy is greater the more orthorexic traits the subjects exhibit.
* Hypothesis 3: The more orthorexic traits subjects exhibit, the more stable they respond (i.e., they respond in the same way to each repetition of the same stimulus) when it comes to categorizing a food as good or bad for health.
* Hypothesis 4: The more severe the orthorexia behaviors, the more distressing the patients will express about their T1D.

ELIGIBILITY:
Inclusion Criteria:

* Person living with type 1 diabetes
* French speaking
* Between 18 and 35 years old

Exclusion Criteria:

* None

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This retrospective study will include data from people living with type I diabetes who participated in the baseline phase of the BETTER registry.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Forced food categorization task according to the categories "healthy / unhealthy" | Baseline
  Instruction to the participant: "Classify the food that appears on your screen as quickly as possible, either as "healthy" (key E) or "unhealthy" (key I).
  Each response and the associated reaction time will be recorded. Stimuli must be classified by the participant as quickly as possible, if the stimulus is not classified before 3 sec the participant moves to the next observation and the stimulus is recorded as NC (not classified).

SECONDARY OUTCOMES:
Stroop Task | Baseline
  Task aimed at evaluating the participant's inhibition and selective attention abilities.
Trail Making Test (TMT) | Baseline
  Task to assess the participant's cognitive flexibility.
Age | Baseline
  In years.
Gender | Baseline
Weight | Baseline
  In kg.
Height | Baseline
  In meters.
Diabetes Information : Age of appearance and duration | Baseline
  In years.
Diabetes Information : How insulin is administered | Baseline
  Pumps or injections.
Diabetes Information : Total dose of insulin | Baseline
  For one day.
Diabetes Information : Duration of diabetes self-monitoring | Baseline
  Number of years or months of its use, either self-monitoring with capillary glucose tests or CGMS, if so.
Diabetes Information : Severe hypoglycemic episodes | Baseline
  Number of severe hypoglycemic episodes over the last year.
Diabetes Information : Diabetes complications | Baseline
  Number and type of diabetes complications.
Eating Habit Questionnaire (EHQ) | Baseline
  Questionnaires for the detection of orthorexic traits.
  Individual subscale and total scale scores are summed, with higher scores indicating increased orthorexia nervosa tendencies.
  The minimum score is 0 and the maximum score is 48.
Ortho-15 Questionnaire | Baseline
  Questionnaires for the detection of orthorexic traits.
  The total score is obtained by adding the scores on each item. A low score on this tool indicates orthorexic tendencies.
  The minimum score is 16 and the maximum is 39.
Eating Disorder Examination Questionnaire (EDE-Q) | Baseline
  Questionnaire for the detection of eating disorders.
  The EDE-Q generates two types of data: frequency data on key behavioural features of eating disorders in terms of number of episodes of the behaviour, and subscale scores reflecting the severity of characteristics of eating disorders.Higher scores on the global scale and subscales denote more problematic eating behaviours and attitudes.
  The minimum score is 0 and the maximum score is 6 for the subscales and the overall scale.
Type 1 Diabetes Distress Scale (T1-DDS) | Baseline
  Questionnaire for the assessment of type 1 diabetes distress.
  The scale yields an overall distress score based on average responses along the 1-6 scale for all 28 items (range = 1-6).
  The scale also yields a score for each of 7 subscales based on the average response on all of the items in that subscale (range = 1-6).
  The higher the score, the higher the distress.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Iceta, MD, PhD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec (IUCPQ)
Locations (2):
- Canada (2):
  - Centre d'expertise Poids, Image et Alimentation (CEPIA), Québec
  - IUCPQ, Québec

IPD SHARING:
Plan to Share IPD: Undecided